CLINICAL TRIAL: NCT03511014
Title: Efficacy of Microcurrent Therapy for Treatment of Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: Elon University, Department of Physical Therapy Education (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HI794-0001
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Acute Knee Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- microcurrent (Experimental)
  Interventions: Device: Microcurrent
- control (Sham Comparator)
  Interventions: Device: Microcurrent

INTERVENTIONS:
Device: Microcurrent — Micrucurrent will be apply

SUMMARY:
The purpose of this study is to evaluate the effect of microcurrent therapy at the knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Pain perceived as a minimum of 3/10 on a 0-10 pain scale
* No phobia of electrical stimulation
* No pain or anti-inflammatory medication will be taken during study
* Injury that began prior to 6-weeks ago before the onset of pain
* Grade II soft tissue injury

Exclusion Criteria:

* Pregnancy
* Diabetes Mellitus
* Neuropathy
* Smoker
* Uncontrolled HTN
* Past surgery in the region to be treated by microcurrent
* Arthritis (RA) in the area to be treated by microcurrent
* Cardiovascular disease
* Allergic to tape/electrodes
* Ligament injury
* Patella Femoral Pain Syndrome (Anterior knee pain)
* Dementia
* Grade III soft tissue injury

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain scale (NRS) for pain (0-10) | 4weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Omron healthcare Co.,Ltd., Mukō, Japan